CLINICAL TRIAL: NCT00786617
Title: The Efficacy of Nurse-driven, Protocol Guided Ventilator Weaning in a Medical-Surgical ICU
Brief Title: The Efficacy of Nurse-driven, Protocol Guided Ventilator Weaning in a Medical-Surgical Intensive Care Unit (ICU)
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-122
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Vent Weaning in Medical- Surgical ICUs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Nurse-driven: Mechanically ventilated patients weaned by nurse-driven ventilator weaning protocol
- Physician-initated: Mechanically ventilated patients weaned by physician-initiated, non-protocol methods

SUMMARY:
1. Mechanically ventilated patients weaned by nurse-driven ventilator weaning protocol will have a mean length of stay on ventilator at least one day shorter than patients weaned by physician-initiated, non-protocol methods
2. Mechanically ventilated patients weaned by nurse-driven ventilator weaning protocol will have al least similar Ventilator, ICU, and Hospital Length Of Stay (LOS) compared to patients weaned by physician-initiated, non-protocol method
3. Nurse-driven ventilator weaning protocol is well accepted by other services: physicians, nurses, and respiratory therapists.

DETAILED DESCRIPTION:
Ventilatory support is one of the most common indications for admission to ICU (1).

The duration of mechanical ventilation is associated with several serious complications, increase mortality, prolong ICU stay, and increase hospital cost (7,8).

Traditionally, the process of ventilator weaning is initiated and carried out my physicians.

Recently, there have been few studies that supported the utility of protocol guided weaning algorithms. Its use have been associated with earlier initiation of weaning, leading to shorter ventilator time, and a trend for shorter ICU length-of-stay and lower hospital costs (1,2,4,9) Several studies have also shown the relative safety of utilizing nursing (3) and RT staff alone or in cooperation with medical staff in the weaning of patients from mechanical ventilation (1,2,6).

We recently developed a nurse-driven ventilator weaning protocol for all ICUs at St. Luke's and Roosevelt hospitals. The protocol was approved by the Critical Care Committee and is implemented as of May 2007. All ICU nurses, respiratory therapists, and ICU physicians have been educated on this protocol We plan to prospectively collect data to look at length of stay on mechanical ventilation in patients weaned by nurse-driven ventilator weaning protocol. We plan to compare such data to retrospectively collected ventilator LOS data in patients weaned by physician-initiated ventilator weaning method.

ELIGIBILITY:
Inclusion Criteria:

* Receiving MV for at least 24 hours in the ICU
* Meeting established protocol criteria for a vent wean trial

Exclusion Criteria:

* Patients in whom MV was actively withdrawn for terminal wean
* Brain dead patients on MV
* Age <18 years old
* Transfers from other hospitals or health care facility who were ventilator dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically Ventilated Patients in Medical-Surgical ICU
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Average Length of Stay on Ventilator | up to 5 months

SECONDARY OUTCOMES:
ICU mortality | up to 5 months
Hospital mortality | up to 5 months
Treatment intensity and resource allocation: Cost of ICU care per year | up to 5 months
Level of acceptance of nurse-driven vent weaning protocol | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Khouli, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center

REFERENCES:
- [Background] Kollef MH, Shapiro SD, Silver P, St John RE, Prentice D, Sauer S, Ahrens TS, Shannon W, Baker-Clinkscale D. A randomized, controlled trial of protocol-directed versus physician-directed weaning from mechanical ventilation. Crit Care Med. 1997 Apr;25(4):567-74. doi: 10.1097/00003246-199704000-00004. PMID 9142019
- [Background] Thorens JB, Kaelin RM, Jolliet P, Chevrolet JC. Influence of the quality of nursing on the duration of weaning from mechanical ventilation in patients with chronic obstructive pulmonary disease. Crit Care Med. 1995 Nov;23(11):1807-15. doi: 10.1097/00003246-199511000-00004. PMID 7587255
- [Background] Ramachandran V, Grap MJ, Sessler CN. Protocol-directed weaning: a process of continuous performance improvement. Crit Care. 2005 Apr;9(2):138-40. doi: 10.1186/cc3053. Epub 2005 Jan 28. PMID 15774063
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Marelich GP, Murin S, Battistella F, Inciardi J, Vierra T, Roby M. Protocol weaning of mechanical ventilation in medical and surgical patients by respiratory care practitioners and nurses: effect on weaning time and incidence of ventilator-associated pneumonia. Chest. 2000 Aug;118(2):459-67. doi: 10.1378/chest.118.2.459. PMID 10936141
- [Background] Salam A, Tilluckdharry L, Amoateng-Adjepong Y, Manthous CA. Neurologic status, cough, secretions and extubation outcomes. Intensive Care Med. 2004 Jul;30(7):1334-9. doi: 10.1007/s00134-004-2231-7. Epub 2004 Mar 4. PMID 14999444
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Dries DJ, McGonigal MD, Malian MS, Bor BJ, Sullivan C. Protocol-driven ventilator weaning reduces use of mechanical ventilation, rate of early reintubation, and ventilator-associated pneumonia. J Trauma. 2004 May;56(5):943-51; discussion 951-2. doi: 10.1097/01.ta.0000124462.61495.45. PMID 15179231
- [Background] Wood G, MacLeod B, Moffatt S. Weaning from mechanical ventilation: physician-directed vs a respiratory-therapist-directed protocol. Respir Care. 1995 Mar;40(3):219-24. PMID 10141679